CLINICAL TRIAL: NCT00749554
Title: Blinded Randomised Placebo-Controlled Trial of TransDiscal Biacuplasty for Patients With Mechanical Low Back Pain of Disc Origin
Brief Title: Trial of Disc Biacuplasty to Treat Chronic Discogenic Low Back Pain
Acronym: TD-RCT-002
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary Investigator Retired.
Sponsor: Baylis Medical Company (Industry)
Collaborators: University of Alberta (Other)
Responsible Party: Dr. Robert S. Burnham, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TD-RCT-Burnham
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Low Back Pain
Keywords: Cooled Radiofrequency; Disc biacuplasty; TransDiscal system; Discogenic pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disc biacuplasty (Active Comparator)
  Interventions: Device: Disc biacuplasty
- Sham treatment. (Placebo Comparator)
  Interventions: Device: Sham biacuplasty

INTERVENTIONS:
Device: Disc biacuplasty — The lesion duration will be 15 minutes with a ramp rate of 2°C per minute and a peak set temperature of 45°C (Temperature in posterior annulus of disc reaches 65°C).
  Other Names: TransDiscal; Cooled Radiofrequency; Intradiscal biacuplasty
  Arms: Disc biacuplasty
Device: Sham biacuplasty — Probes not inserted into disc, no RF electricity applied.
  Arms: Sham treatment.

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the effectiveness of Disc Biacuplasty in relieving pain, reducing medication intake and improving function, satisfaction and quality of life of patients with chronic mechanical discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Able to understand the informed consent and baseline/follow-up questionnaires
* Chronic low back pain > leg pain for longer than 6 months, unresponsive to comprehensive non-operative treatment
* No clinical evidence of SI joint mediated pain
* Concordant pain reproduced on provocative discography at an intensity of >6/10 at low pressure (<50 psi) at not more than 2 discs and a negative response at an adjacent control disc
* Preservation of at least 50% height of the symptomatic disc(s)

Exclusion Criteria:

* Active radicular pain
* Nucleus pulposus herniation > 5 mm, extrusion or sequestration on MRI
* Spondylolithesis at the symptomatic level
* Prior surgery at the symptomatic level
* Concomitant cervical or thoracic pain >2/10 (VAS) in severity
* Other chronic pain conditions (i.e. Fibromyalgia Syndrome)
* Immunosuppression (i.e. Cancer, AIDS, Rheumatoid arthritis)
* Third-party (WSIB, litigation or insurance) involvement
* Psychological issues impeding recovery by history, examination and/or a Beck Depression Inventory score of >20
* Systemic or localized infection (at the anticipated needle entry sites)
* BMI > 35 (Obesity)
* Substance or opioid abuse
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Duration (months) of greater than 50% pain relief compared to pre-procedure baseline on the visual analogue scale (VAS). | 12 months

SECONDARY OUTCOMES:
Oswestry Disability Index | 12 months
Assessment of Quality of Life | 12 months
SF-36 for physical functioning | 12 months
Reduction in Medication Intake | 12 months
Patient satisfaction | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Burnham, MD, Principal Investigator — University of Alberta
Locations (1):
- Lacombe Hospital, Lacombe, Alberta, Canada

REFERENCES:
- [Background] Kapural L, Ng A, Dalton J, Mascha E, Kapural M, de la Garza M, Mekhail N. Intervertebral disc biacuplasty for the treatment of lumbar discogenic pain: results of a six-month follow-up. Pain Med. 2008 Jan-Feb;9(1):60-7. doi: 10.1111/j.1526-4637.2007.00407.x. PMID 18254768
- [Background] Kapural L. Intervertebral disk cooled bipolar radiofrequency (intradiskal biacuplasty) for the treatment of lumbar diskogenic pain: a 12-month follow-up of the pilot study. Pain Med. 2008 May-Jun;9(4):407-8. doi: 10.1111/j.1526-4637.2008.00464.x. No abstract available. PMID 18489632